CLINICAL TRIAL: NCT03990532
Title: Phase I/II Dose Escalation by Simultaneous Integrated Boost for Mediastinal Lymph Node Recurrence After Radical Surgery of Esophageal Cancer
Brief Title: Simultaneous Integrated Boost for Mediastinal Lymph Node Recurrence After Radical Surgery of Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shengguang Zhao, associate chief physician, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH2019-69
Record Dates: First submitted 2019-06-16; First posted 2019-06-19 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Cancer; Salvage Radiotherapy; Dose-escalation; Mediastinal Lymph Node Recurrence
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Radiation: treatment group(phase I); Radiation: treatment group (phase II)

INTERVENTIONS:
Radiation: treatment group(phase I) — Dose-escalation plan (phase I)
  Radiotherapy:
  LEVEL 1: dose given at PTV-G will be 58.8Gy/28 fractions； 2.1Gy/per fraction; LEVEL 2: dose given at PTV-G will be 64.4Gy/28 fractions； 2.3Gy/per fraction; LEVEL 3: dose given at PTV-G will be 70Gy/28 fractions； 2.5Gy/per fraction Concurrent chemotherapy: 5-Fu/capecitabine/S-1+DDP or S-1 or Capecitabine
Radiation: treatment group (phase II) — Radiotherapy dose was prescribed according to phase I trial results; Concurrent chemotherapy: 5-Fu/capecitabine/S-1+DDP or S-1 or Capecitabine

SUMMARY:
Esophageal cancer (EC) ranks the seventh most diagnosed malignant tumor (572,000 new cases) and the sixth cancer-related mortality (509,000 deaths) worldwide in 2018. The incidence of EC is strikingly varying among the regions and sexes. Approximately 70% of EC cases occur in men, and there is a 2-fold to 3-fold difference in incidence and mortality rates between regions worldwide. According to the latest reported in 2017, esophageal cancer ranks the sixth most common cancer and the fourth leading cause of cancer-mortality in China. Currently, esophagectomy is considered as the standard treatment for resectable EC patients. However, the prognosis of stage IIA-III esophageal cancer after esophagectomy remains poor, and local regional lymph node recurrence is the major patterns of recurrence, and mediastinal lymph node recurrence is one of the most common sites. Previous retrospective study has found that salvage chemoradiotherapy is a effective treatment option for these patients. However, the optimal dose remains unknown. In addition, no prospective trials have been conducted to investigate the efficacy and toxicities of salvage chemo-radiotherapy by using simultaneous integrated boost for the treatment of mediastinal lymph node recurrence after radical surgery of esophageal Cancer

ELIGIBILITY:
Inclusion Criteria:

Histo-pathologically proven diagnosis of esophageal squamous cell carcinoma. Age ≥18 and ≤80 ECOG performance status 0-1. Clinical diagnosis of ≤5 mediastinal lymph nodes recurrence after esophagectomy.

Patients without distant metastasis and life expectancy ≥ 3 months. adequate liver and renal function and adequate bone marrow reservation. Written, signed informed consent.

Exclusion Criteria:

Prior radiotherapy to recurrence site of esophageal cancer. Other co-existing malignancies or malignancies diagnosed within the last 5 years.

Pregnant women. Women who are breastfeeding a baby. Patients with uncontrolled serious medical or mental illnesses.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity(DLT) of Simulatianeous Integrated Boost (SIB) | up to 3 months
  DLT was defined as grade 4 or higher hematological toxicities and/or grade 3 or higher nonhematological toxicities.
Overall survival (phase II) | up to 1 year
  Survival time was measured from the date of study enrollment to the date of death or last follow-up;

SECONDARY OUTCOMES:
Overall survival (phase I) | up to 1 year
  Survival time was measured from the date of study enrollment to the date of death or last follow-up;
Late toxicity (phase I) | up to 2 year
  late toxicity were grade according to RTOG and CTCAE criteria
Overall survival (phase II) | up to 2 year
  Survival time was measured from the date of study enrollment to the date of death or last follow-up;
acute Toxicity (phase II) | up to 3 months
  acute toxicity were grade according to CTCAE criteria
late Toxicity (phase II) | up to 2 year
  late toxicity were grade according to RTOG and CTCAE criteria
1-year local progression-free survival | up to 1 year
  From treatment initiation to first documented local progression or death or censor

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China